CLINICAL TRIAL: NCT02938143
Title: Progressive Tendon-loading Exercise Therapy for Patellar Tendinopathy in Jumping Athletes: A Randomized Controlled Clinical Trial Evaluated With Advanced 3D UTE MR
Brief Title: Exercise Therapy for Patellar Tendinopathy Evaluated With Advanced UTE-MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Edwin Oei, dr, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTE MRI
Record Dates: First submitted 2016-10-03; First posted 2016-10-19 (Estimated); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Tendinopathy
Keywords: Jumpers knee; Patellar Tendinopathy; Jumping Athletes; UTE MRI; Exercise Therapy; NBA
MeSH Terms: conditions — Tendinopathy | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4-stage criteria-based exercise protocol (Experimental): a progressive 4-stage criteria-based exercise protocol within the limits of pain
  Interventions: Procedure: Exercise
- Heavy-load eccentric exercise protocol (Active Comparator): a 12-week painful heavy-load eccentric exercise protocol
  Interventions: Procedure: Exercise (usual care)

INTERVENTIONS:
Procedure: Exercise — The intervention treatment is a progressive 4-stage criteria-based exercise protocol within the limits of pain, consisting of progressive isometric, isotonic, plyometric, and sport-specific exercises.24 Progression criteria are individualized.
  Arms: 4-stage criteria-based exercise protocol
Procedure: Exercise (usual care) — The control treatment is a painful heavy-load eccentric exercise program performed twice daily with 3 sets of 15 repetitions for 12 weeks on a 25° decline board. The downward component (eccentric component) will be performed with the symptomatic leg and the upward component (concentric phase) on the asymptomatic leg.
  Arms: Heavy-load eccentric exercise protocol

SUMMARY:
Patellar tendinopathy is a frequent overuse injury that causes pain and impaired performance in jumping athletes. Exercise therapy is considered the best initial treatment option for tendinopathies as clinical improvements in pain and function have been demonstrated. Although painful eccentric exercise protocols have been promoted as standard care based on positive results in early studies, a recent systematic review demonstrated that these are not associated with improved tendon structure and are ineffective when applied in-season. Progressive tendon-loading exercise therapy for patellar tendinopathy constitutes a novel concept in sports medicine. A recent study advocates a progressive 4-stage criteria-based exercise protocol as it results in a less reactive tendon and ability to restore collagen alignment. This protocol consists of progressive isometric, isotonic, plyometric, and sport-specific exercises. Isometric exercises have been shown to reduce pain and decrease motor cortex inhibition of the quadriceps. This approach would enable jumping athletes to resume sports within the limits of pain, with improved muscle function, and sufficient tendon structure re-organization. The diagnostic imaging work-up of patellar tendinopathy typically consists of ultrasound, magnetic resonance imaging (MRI), or a combination of both. Ultrashort echo time (UTE) MRI is an advanced MRI technique, which enables assessment of tissues with short T2-time, such as tendon, the structure of which is invisible on regular MRI. UTE has been shown to quantitatively depict changes in tendon microstructure and therefore allows in-vivo evaluation of tendon regeneration. It is currently unknown whether quantitative UTE MRI parameters change after exercise treatment, are related to clinical symptoms of patellar tendinopathy, have prognostic value for exercise treatment response, and offer additional value over ultrasound

DETAILED DESCRIPTION:
Patellar tendinopathy ('jumper's knee') is a clinical condition of gradually progressive activity-related pain at the insertion of the patellar tendon at the apex patellae. Prolonged repetitive stress of the knee-extensor apparatus can lead to this common overuse tendinopathy in athletes from different sports, resulting in pain and impaired performance in athletes. High prevalence rates have been reported in jumping sports such as volleyball and basketball (45% and 32% in elite athletes, respectively). Symptoms can be long-standing if not treated appropriately in the initial stages. Furthermore, there is currently no strong evidence for second-line treatments such as shockwave therapy and platelet-rich plasma. Therefore, it is important to improve exercise protocols as a first treatment of choice.

Tendinopathy is a widely accepted, generic term that encompasses any abnormal condition of a tendon. Clinical symptoms include activity-related pain associated with tenderness, localized swelling and impaired performance. Histopathologically, tendinopathy is characterized by structural disorganization of the tendon collagen that alters the loading capacity of a specific tendon.

Exercise therapy is considered as the best initial treatment option for tendinopathies as histopathological changes and clinical improvements on pain and function have been demonstrated. Most studies have been conducted using eccentric exercise protocols and early studies showed positive effects, resulting in promoting these isolated painful exercises as standard care. One hypothesis behind the potential beneficial effects of eccentric exercises is that increased load results in increased collagen synthesis and subsequent healing response. However, a recent systematic review demonstrated that the available literature does not support observable structural change as an explanation for the response of eccentric exercises. Furthermore, eccentric exercises may not be effective for reducing pain and improving strength when used in-season and might even increase symptoms in jumping athletes with patellar tendon pathology.

Progressive tendon-loading exercise therapy for patellar tendinopathy constitutes a novel concept in sports medicine. A recent publication advocates a progressive 4-stage criteria-based exercise protocol within the limits of pain, consisting of progressive isometric, isotonic, plyometric, and sport-specific exercises, resulting in a less reactive tendon, immediate decreased pain levels, diminished motor cortex inhibition of the quadriceps muscles, and potential to restore collagen alignment. These new insights are completely conflicting with the painful heavy-load eccentric exercise protocols currently applied as usual care. It is currently unknown which exercise therapy is the best strategy for athletes with patellar tendinopathy, as adequately powered randomized studies are lacking.

Although clinical examination represents the gold standard in the diagnosis of patellar tendinopathy, it is commonplace to perform diagnostic imaging of the patellar tendon to confirm the diagnosis and rule out alternative diagnoses. Furthermore, imaging can be used to estimate response to treatment. This diagnostic imaging work-up usually consists of magnetic resonance imaging (MRI), ultrasound or, occasionally, a combination of both. On "regular" MRI, increased tendon size and visually increased signal intensity within the proximal patellar tendon can be observed in patellar tendinopathy , but altered tendon microstructure is invisible. A novel innovative method to detect tendon abnormalities is the ultrashort echo time (UTE) MRI technique. UTE enables accurate detection of changes in a reactive tendon both visually and in a quantitative manner by measuring T2* relaxation time UTE MRI has also been shown to quantitatively depict changes in tendon microstructure and, therefore, this innovative imaging modality allows in-vivo evaluation of tendon regeneration. It is currently unknown whether quantitative UTE MRI parameters change after exercise treatment, are related to clinical symptoms of patellar tendinopathy, and have prognostic value for exercise treatment response.

ELIGIBILITY:
Inclusion Criteria:

Age 18-35 years old (the chosen age range will minimize chances of other conditions causing anterior knee pain such as osteoarthritis and osteochondrotic diseases like Sinding-Larsen-Johansson syndrome and Osgood-Schlatter disease) History of knee pain in patellar tendon or its patellar or tibial insertion in association with training and competition Playing sports for at least 3 times a week Palpation tenderness to the corresponding painful area On ultrasound, there needs to be a fusiform tendon thickening and/or decreased tendons structure and/or increased Doppler signal within the patellar tendon27 VISA-P score < 80/100 points

Exclusion Criteria:

Known presence of inflammatory joint diseases (e.g. spondylarthropathy, gout or rheumatoid arthritis) or familial hypercholesterolaemia.

Contraindications for MRI (pregnancy, metallic implants, etc.) Daily use of drugs with a putative effect on the patellar tendon in the preceding year (e.g. fluoroqinolones and statins) Knee surgery in the history of the index knee Previous patellar tendon rupture of the index knee Local injection therapy with corticosteroids in the preceding 12 months Daily exercise therapy with a minimum duration of 4 weeks in total in the preceding 12 months Acute knee or patellar tendon injuries Inability to perform an exercise program Participation in other concomitant treatment programs Signs or symptoms of other coexisting knee pathology on physical examination (such as joint effusion and joint line tenderness) or additional diagnostics (Chondral lesion of the patella or trochlea on MRI or prepatellar bursitis on US).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The change of the validated and disease-specific VISA-P score over 24 weeks | 24 weeks
  The change of the validated and disease-specific VISA-P score over 24 weeks

SECONDARY OUTCOMES:
Subjective patient satisfaction | 3 years
  Subjective patient satisfaction (excellent / good / fair / poor)
Return to sports | 3 years
  Return to sports (Return to desired sport on pre-injury level / return to desired sport but on a lower level / return to sports but not desired sport / no return to sports
Time to return to full training in desired sport | 3 years
  Time to return to full training in desired sport
Pain rating on a Visual Analogue Scale (VAS) | 3 years
  Pain rating on a Visual Analogue Scale (VAS) in which 0 represents no pain, and 100 maximal pain
Strength (N.kg.m) of the abductors and quadriceps muscles using dynamometry | 3 years
  Strength (N.kg.m) of the abductors and quadriceps muscles using dynamometry Leg length of the upper extremity will be measured to be able to correct for lever arm.
Flexibility of the calf muscles using the weight-bearing dorsiflexion lunge tes | 3 years
  Flexibility of the calf muscles using the weight-bearing dorsiflexion lunge tes
Compliance to the exercise program (total percentage of prescribed exercises performed). | 3 years
  Compliance to the exercise program (total percentage of prescribed exercises performed). This will be asked on a weekly basis using a short online questionnaire.
Training load | 3 years
  Training load, which is defined as: Total duration of training and match play per week (minutes) multiplied by the experienced intensity of training sessions and games using the modified Borg CR-10 RPE scale.46 This will be asked on a weekly basis using a short online questionnaire.
MRI: Conventional: maximum anterior-posterior (AP) thickness and signal abnormalities | 3 years
  Conventional: maximum anterior-posterior (AP) thickness and signal abnormalities (intratendinous, peritendinous).
MRI: 3D UTE Cones: T2* relaxation time | 3 years
  3D UTE Cones: T2* relaxation time

OTHER OUTCOMES:
US:· Grey scale: maximum anterior-posterior (AP) thickness, presence of calcification | 3 years
  Grey scale: maximum anterior-posterior (AP) thickness, presence of calcification
US: PDU: Doppler signal (neovascularisation score determined with the modified Ohberg Scale). | 3 years
  PDU: Doppler signal (neovascularisation score determined with the modified Ohberg Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Edwin H Oei, Dr, Principal Investigator — Erasmus Medical Center; Robert-Jan de Vos, Dr., Principal Investigator — Erasmus Medical Center; S Breda, Drs., Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deng J, Breda SJ, Eygendaal D, Oei EH, de Vos RJ. Association Between Physical Tests and Patients-Reported Outcomes in Athletes Performing Exercise Therapy for Patellar Tendinopathy: A Secondary Analysis of the JUMPER Study. Am J Sports Med. 2023 Nov;51(13):3523-3532. doi: 10.1177/03635465231200241. Epub 2023 Oct 10. PMID 37815096

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT02938143/SAP_000.pdf